CLINICAL TRIAL: NCT00268385
Title: A Phase I Study of Vorinostat (Suberoylanilide Hydroxamic Acid [SAHA]) in Combination With Temozolomide in Patients With Malignant Gliomas
Brief Title: Vorinostat and Temozolomide in Treating Patients With Malignant Gliomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00675; NCI-2009-00675 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NABTC 04-03; CDR0000450762; NABTC04-03 (Other: Adult Brain Tumor Consortium); NABTC-04-03 (Other: CTEP); U01CA137443 (NIH); U01CA062399 (NIH)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Temozolomide; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vorinostat, temozolomide) (Experimental): PART I: Patients receive vorinostat PO QD or BID on days 1-7 and 15-21 OR QD or BID on days 1-7. Patients also receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Treatment may continue beyond 13 courses at the discretion of the investigator.
  PART II: Patients receive vorinostat and temozolomide as in part I*.
  [Note: Beginning in course 2, some patients may receive a higher dose of temozolomide.]
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temozolomide; Drug: Vorinostat

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temozolomide — Given orally
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Drug: Vorinostat — Given orally
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with temozolomide in treating patients with malignant gliomas. Drugs used in chemotherapy, such as vorinostat and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vorinostat may help temozolomide work better by making tumor cells more sensitive to the drug. Giving vorinostat together with temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of vorinostat (suberoylanilide hydroxamic acid [SAHA]) in combination with temozolomide in patients with malignant gliomas.

II. To characterize the safety profile of vorinostat (SAHA) in combination with temozolomide.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of vorinostat (SAHA) in combination with temozolomide.

II. To determine efficacy of vorinostat (SAHA) in combination with temozolomide as measured by objective response.

TERTIARY OBJECTIVES:

I. To explore the association of response to treatment to the molecular phenotype of the tumor.

II. To assess the effects of vorinostat (SAHA) on histone acetylation status in peripheral mononuclear cells.

OUTLINE: This is a 2-part, dose-escalation study of vorinostat.

PART I: Patients receive vorinostat orally (PO) once (QD) or twice daily (BID) on days 1-7 and 15-21 OR QD or BID on days 1-7. Patients also receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Beginning in course 2, some patients may receive a higher dose of temozolomide. Treatment may continue beyond 13 courses at the discretion of the investigator.

PART II: Patients receive vorinostat and temozolomide as in part 1*.

[Note: *Beginning in course 2, all patients receive a higher dose of temozolomide.]

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven intracranial malignant glioma will be eligible for this protocol; malignant gliomas include glioblastoma multiforme (GBM), gliosarcoma (GS), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified); patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a malignant glioma is made
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must have signed an authorization for the release of their protected health information; patients must be registered with the Adult Brain Tumor Consortium (ABTC) Central Office database prior to treatment with study drug
* Life expectancy > 8 weeks
* Karnofsky performance status of >= 60
* White blood cell (WBC) >= 3,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL; eligibility level for hemoglobin may be reached by transfusion
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* If liver function tests are above the institutional upper limit of normal but < 2 times institutional upper limit of normal, the decision to initiate temozolomide treatment should carefully consider the benefits and risks for the individual patient
* Creatinine < 1.5 mg/dL
* A scan should be performed within 14 days prior to registration and on a steroid dose that has been stable for at least 5 days; if the steroid dose is increased between the date of imaging and registration a new baseline magnetic resonance (MR)/computed tomography (CT) is required; the same type of scan, i.e., magnetic resonance imaging (MRI) or CT must be used throughout the period of protocol treatment for tumor measurement
* Patients must have an interval of greater than or equal to 3 weeks (21) days from the completion of radiation therapy to study entry
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 7 days prior to registration; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of participation in the study
* Patients must be willing to participate in the pharmacokinetic studies
* ELIGIBILITY CRITERIA SPECIFIC FOR PATIENTS IN PART I OF THE STUDY
* Patients with either stable disease after radiation therapy or with progression are eligible (except if they have progressed on temozolomide; patients who have received prior treatment with temozolomide and have stable disease are eligible
* Patients with recurrent disease may have had treatment for any number of prior relapses; relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy)
* Patients must have recovered from the toxic effects of prior therapy: 28 days from any investigational agent, 28 days from prior cytotoxic therapy except 23 days from last dose of temozolomide for patients taking the standard 5 days every 28 day regimen of temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration, and 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count); any questions related to the definition of non-cytotoxic agents should be directed to the study chair
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * They have recovered from the effects of surgery
  * Residual disease following resection is not mandated for eligibility into the study; to best assess the extent of residual disease post-operatively, a CT/MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to registration; if the 96-hour scan is more than 14 days before registration, the scan needs to be repeated; if the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or thallium scanning, MR spectroscopy or surgical documentation of disease
* ELIGIBILITY CRITERIA SPECIFIC FOR PATIENTS IN PART II OF THE STUDY
* Only patients with stable disease after radiation therapy are eligible for part 2 of the study; patients with recurrent disease are ineligible
* The only prior therapy permitted for patients in part 2 of the study is concomitant temozolomide with radiation therapy or radiation therapy alone; patients that are stable on adjuvant temozolomide may also participate
* Patients with recurrent disease and prior chemotherapies (except concurrent or adjuvant temozolomide) will not be included in this part of the study

Exclusion Criteria:

* Patients who have progressed on temozolomide are ineligible
* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* Patients must not have active infection or serious intercurrent medical illness
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat (SAHA); potential risks may also apply to temozolomide
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism
* Patients who are known to be human immunodeficiency virus (HIV) positive and are receiving combination antiretroviral therapy are ineligible
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA) or other agents used in study
* Patients should not have taken valproic acid (another histone deacetylase inhibitor) for at least 2 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-12-16 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
MTD of vorinostat with temozolomide defined as the dose at which less than one-third of patients experience dose-limiting toxicity based on the CTC severity grading (Part I) | 28 days
  For both parts of the study, treatment administration will be described for all cycles. Doses administered, dose modifications/delays, and duration of therapy will be evaluated. Safety variables summarized by descriptive statistics. Adverse events that occur will be reported for each dose level and described in terms of incidence and severity. Laboratory data will be presented by dose level at each observation time. Values outside of normal limits will be identified and their frequency calculated. Distribution by CTC severity grade (when applicable) and clinical relevance will be given.

SECONDARY OUTCOMES:
Efficacy in terms of anti-tumor activity based on clinical, radiographic, and biologic assessments (Part II) | Up to 4 years
  A descriptive analysis of evidence of anti-tumor activity will be provided based on clinical, radiographic, and biologic assessments of efficacy.
Plasma pharmacokinetic parameters of vorinostat | Baseline, 1, 2, 3, 4, 6, 8, and 24 hours post-dose day 1 of course 1
  Presented in tabular and graphic form. Pharmacokinetic parameters of interest such as maximal plasma concentration (Cmax), time of maximal concentration (Tmax), area under the plasma concentration-time curve (AUCo-t and AUC-infinity), clearance (CL), apparent volume of distribution at steady state (Vdss), terminal half-life (t1/2), and tumor to plasma (whole blood) concentration ratio will be determined using non-compartmental methods. Dose proportionality in pharmacokinetic parameters will be determined by performing a one-way analysis of variance (ANOVA) on dose-normalized parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, Principal Investigator — National Cancer Institute (NCI)
Locations (17):
- United States (17):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin